CLINICAL TRIAL: NCT07269717
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial on the Efficacy and Safety of HRS-1893 in the Treatment of Heart Failure With Preserved Ejection Fraction
Brief Title: A Phase II Clinical Trial of HRS-1893 in the Treatment of Heart Failure With Preserved Ejection Fraction
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRS-1893-203
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-1893 Tablet Group (Experimental)
  Interventions: Drug: HRS-1893 Tablet
- HRS-1893 Tablet Placebo Group (Placebo Comparator)
  Interventions: Drug: HRS-1893 Tablet Placebo

INTERVENTIONS:
Drug: HRS-1893 Tablet — HRS-1893 tablet.
  Arms: HRS-1893 Tablet Group
Drug: HRS-1893 Tablet Placebo — HRS-1893 tablet placebo.
  Arms: HRS-1893 Tablet Placebo Group

SUMMARY:
This study aims to evaluate the safety and tolerability of HRS-1893 in subjects with heart failure with preserved ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years at screening, regardless of gender;
2. Body mass index < 35 kg/m²;
3. Diagnosed with chronic heart failure before screening, and meeting relevant diagnostic criteria during the screening period: (1) Transthoracic echocardiography (TTE) at screening showing a resting left ventricular ejection fraction (LVEF) ≥ 60%; (2) Elevated N-terminal pro-B-type natriuretic peptide (NT-proBNP) during the screening period; (3) Echocardiography showing structural or functional abnormalities of the heart, etc.;
4. New York Heart Association (NYHA) classification of II or III at screening;
5. KCCQ-CSS score between ≥25 and ≤75 at screening;
6. Resting oxygen saturation >90% without supplemental oxygen at screening;
7. Female participants of childbearing potential must have a negative serum pregnancy test before the first dose and must not be breastfeeding during the study. Female participants of childbearing potential and male participants whose partners are women of childbearing potential must agree to avoid donating sperm/eggs from the time of signing the informed consent until three months after the last dose of the study drug and comply with relevant contraceptive requirements;
8. Understand the study procedures and methods, voluntarily participate in this trial, and provide written informed consent.

Exclusion Criteria:

1. Previously diagnosed or found during screening with hypertrophic cardiomyopathy (HCM), or having infiltrative/genetic/storage diseases that cause heart failure with preserved ejection fraction (HFpEF)/myocardial hypertrophy (such as amyloidosis, Fabry disease, Noonan syndrome with left ventricular hypertrophy), or complete M protein or monoclonal light chain (such as κ or λ) detected in serum protein electrophoresis and serum immunofixation electrophoresis during screening (researchers may deem not applicable if amyloidosis/multiple myeloma are excluded);
2. Previously diagnosed or found during screening with hyperthyroidism;
3. At any time in their clinical history, previously experienced left ventricular systolic dysfunction (LVEF <45%);
4. History of syncope or sustained ventricular tachycardia within 6 months prior to screening;
5. Previously experienced cardiac arrest with resuscitation at any time or received ICD therapy for life-threatening ventricular arrhythmia within 6 months prior to screening;
6. Previously diagnosed or found during screening with atrial fibrillation;
7. Coronary artery disease (stenosis >70% in one or more coronary arteries) or myocardial infarction: newly developed within 6 months prior to screening, or occurred more than 6 months prior without completed revascularization (such as percutaneous coronary intervention or coronary artery bypass grafting);
8. Moderate to severe aortic stenosis, hemodynamically significant mitral stenosis, or severe mitral/tricuspid regurgitation at screening (as determined by the investigator);
9. Severe chronic obstructive pulmonary disease (COPD) or other pulmonary diseases requiring home oxygen therapy, chronic nebulization/oral steroid treatment, or hospitalization due to pulmonary decompensation in the past 12 months;
10. Acute respiratory infection at screening;
11. Required intravenous diuretics, inotropes, vasodilators, or left ventricular assist device therapy for acute decompensated heart failure within 30 days prior to screening;
12. Clinically significant history of malignancy within the past 5 years (excluding cancers that have been confirmed cured or in remission for ≥5 years, basal or squamous cell skin cancer that was radically excised within 5 years, carcinoma in situ of the cervix, and excised colon polyps);
13. Electrocardiogram abnormalities posing safety risks at screening (as determined by the investigator, such as second-degree type II AV block, complete AV block, symptomatic ventricular arrhythmias, torsades de pointes, etc.);
14. Any clinically significant abnormal screening laboratory values during screening deemed unsuitable for enrollment by the investigator;
15. Positive result in any infectious disease screening during screening, including hepatitis B surface antigen, hepatitis C antibody, syphilis antibody, HIV antibody (or AIDS virus antibody or P24 antigen);
16. Inability to complete the six-minute walk test during screening (e.g., due to leg fractures, post-stroke mobility impairment);
17. Patients who received β-blockers, diltiazem, or verapamil prior to screening but were not on a stable dose for more than 4 weeks before randomization, or are expected not to maintain the same medication regimen during the trial;
18. Subjects who received heart failure medication treatment (diuretics, sodium-glucose co-transporter 2 inhibitors [SGLT2i], angiotensin receptor-neprilysin inhibitors [ARNI], mineralocorticoid receptor antagonists [MRA], angiotensin-converting enzyme inhibitors [ACEI], angiotensin II receptor blockers [ARB], glucagon-like peptide-1 [GLP-1] or GLP-1/glucose-dependent insulinotropic polypeptide [GIP]) prior to screening but have not been on a stable dose for more than 4 weeks before randomization, or are expected to be unable to maintain the same medication regimen during the trial;
19. Subjects who used a myosin inhibitor within a period shorter than 5 half-lives before the trial drug administration;
20. Subjects who participated in any drug or medical device clinical trial within 3 months prior to screening (participation in a clinical trial is defined as the subject having received the trial drug or medical device treatment);
21. Other conditions deemed by the investigator that make the subject unsuitable for participation in the trial, such as conditions that may increase trial risk, affect the subject's protocol compliance, or impact the subject's ability to complete the trial due to physiological or psychological diseases or conditions.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs). | Week 24.
  In heart failure patients with preserved ejection fraction after treatment with HRS-1893.

SECONDARY OUTCOMES:
Change from baseline in N-terminal pro B-type natriuretic peptide (NT-proBNP). | Week 12 and Week 24.
  In heart failure patients with preserved ejection fraction after treatment with HRS-1893.
Change from baseline in Kansas City Cardiomyopathy Questionnaire-Clinical Summary Score (KCCQ-CSS). | Week 12 and Week 24.
  In heart failure patients with preserved ejection fraction after treatment with HRS-1893.
Proportion of heart failure patients with preserved ejection fraction with an improvement of ≥1 NYHA functional class from baseline. | Week 12 and Week 24.
  In heart failure patients with preserved ejection fraction after treatment with HRS-1893.
Change from baseline in total distance walked during the six-minute walk test (6MWT). | Week 12 and Week 24.
  In heart failure patients with preserved ejection fraction after treatment with HRS-1893.
Change from baseline in resting left ventricular ejection fraction (LVEF). | Week 12 and Week 24.
  In heart failure patients with preserved ejection fraction after treatment with HRS-1893.
Plasma concentration of HRS-1893. | Up to about 29 weeks.
  In heart failure patients with preserved ejection fraction after treatment with HRS-1893.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided